CLINICAL TRIAL: NCT04745910
Title: Effect of Pegloticase on Reduction of Uric Acid in Patients With Tumor Lysis Syndrome: A Pilot Pragmatic Clinical Trial
Brief Title: Pegloticase for the Reduction of Uric Acid in Patients With Tumor Lysis Syndrome
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0330; NCI-2020-13890 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0330 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Tumor Lysis Syndrome
MeSH Terms: conditions — Hematologic Neoplasms; Tumor Lysis Syndrome | interventions — Pegloticase; Urate Oxidase; Carbamates; Oxidoreductases; Uric Acid; Amides; rasburicase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pegloticase) (Experimental): Patients receive pegloticase IV over 120 minutes. Patients whose serum uric acid does not drop below 6 mg/dL within 24 hours receive a second dose of pegloticase IV over 120 minutes on day 2. Patients whose serum uric acid does not drop below 6 mg/dL after two doses of pegloticase receive standard of care rasburicase IV QD for 5 days.
  Interventions: Drug: Pegloticase; Drug: Rasburicase

INTERVENTIONS:
Drug: Pegloticase — Given IV
  Other Names: Des-(1-6)-(7-threonine,46-threonine,291-lysine,301-serine)uricase (EC 1.7.3.3, urate oxidase) Sus scrofa (pig) tetramer, Non Acetylated, Carbamates with alpha-carboxy-omega-methoxypoly(oxyethylene); Krystexxa; Methoxypolyethylene Glycol Uricase; Oxidase, Urate (Synthetic Sus scrofa variant pigks-DN subunit), homotetramer, amide with alpha-carboxy-omega-methoxypoly(oxy-1,2-ethanediyl); Polyethylene Glycol-uricase; Puricase
Drug: Rasburicase — Given IV
  Other Names: Elitek; Recombinant Urate Oxidase; SR 29142; SR-29142; Urate Oxidase

SUMMARY:
This trial studies the effect of pegloticase in reducing uric acid levels in patients with hyperuricemia (high blood levels of uric acid) caused by tumor lysis syndrome. Tumor lysis syndrome occurs when the breakdown products of cancer cells, such as uric acid, enter the blood stream. High levels of uric acid in blood may cause kidney damage and reduce kidney function. The goal of this trial is to learn if pegloticase may lower uric acid levels in blood when given to cancer patients with hyperuricemia caused by tumor lysis syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To collect preliminary data on the effectiveness of a single dose of pegloticase in lowering serum uric acid levels to less than 6.0 mg/dl within 24 hours in patients with hyperuricemia in the setting of tumor lysis syndrome.

SECONDARY OBJECTIVES:

I. To assess the effect of pegloticase on renal function in patients with hyperuricemia in the setting of tumor lysis syndrome as measured by changes in serum creatinine/estimated glomerular filtration rate (eGFR) and urine output.

II. To estimate the rate of renal replacement therapy initiation for acute kidney injury secondary to tumor lysis syndrome among patients treated with pegloticase.

OUTLINE:

Patients receive pegloticase intravenously (IV) over 120 minutes. Patients whose serum uric acid does not drop below 6 mg/dL within 24 hours receive a second dose of pegloticase IV over 120 minutes on day 2. Patients whose serum uric acid does not drop below 6 mg/dL after two doses of pegloticase receive standard of care rasburicase IV once daily (QD) for 5 days.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfill the following criteria:

1. Signed informed consent prior to any study specific procedures (patient or caregiver)
2. Male or female 18 years of age or older
3. In the investigator's opinion, expected survival of at least 1 month
4. Deemed stable by the investigator
5. Serum Uric Acid ≥ 6 mg/dL
6. Risk for tumor lysis syndrome based on the MD Anderson TLS risk score

Exclusion Criteria:

Patients will be ineligible for study enrollment if any of the following exclusion criteria are fulfilled:

1. Inability or refusal to give informed consent (patient or caregiver)
2. Subject unwilling to take study medication
3. Known allergy to uricase
4. Pregnant
5. Breastfeeding
6. Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
7. Transfusion in last 7 days (as this interferes with G6PD test), with the exception of platelet transfusions.
8. Has received rasburicase during current admission.(Can be considered i24 hours after last Rasburicase administered, current or previous admission)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | Within 24 hours of single dose of pegloticase
  Will estimate the 24-hour response rate along with the corresponding 90% confidence interval. In addition, the report will present plots of uric acid levels across all time points.

SECONDARY OUTCOMES:
Time from pegloticase infusion until serum uric acid levels drop to 6 mg/dL | Up to 14 days after pegloticase administration
  Will display results in frequency tables and plots of serum uric acid levels across time.
Renal function | Up to 14 days after pegloticase administration
  Will summarize serum creatinine and estimated glomerular filtration rate at each time point and plot these lab values across time. Finally, will calculate the rate and 90% confidence interval for the initiation of renal replacement therapy within the 14-day observation window.

OTHER OUTCOMES:
Serum uric acid level | Up to 14 days after pegloticase administration
  Will examine the association of baseline characteristics with serum uric acid level using the Fisher's exact test, student's t-test, paired t-test, Wilcoxon rank-sum test, or Wilcoxon signed-rank test and will employ graphical methods when useful.

CONTACTS AND LOCATIONS:
Overall Officials: Sreedhar Mandayam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org